CLINICAL TRIAL: NCT01024751
Title: A Study to Evaluate the Clinical Performance of a Novel Multipurpose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Mohinder Merchea, OD, PhD, MBA, Bausch & Lomb Incorporated
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 636
Record Dates: First submitted 2009-11-30; First posted 2009-12-03 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-07

CONDITIONS: Ocular Discomfort

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bausch & Lomb Multi-Purpose Solution (Experimental): Multi-Purpose Solution to be used for disinfecting contact lenses.
  Interventions: Device: Bausch & Lomb Multi-Purpose Solution
- Ciba's Multi-Purpose Solution (Active Comparator): Multi-Purpose Solution to be used for disinfecting contact lenses.
  Interventions: Device: Ciba's Multi-Purpose Solution

INTERVENTIONS:
Device: Bausch & Lomb Multi-Purpose Solution — Lens care product for disinfecting lenses on a daily basis.
  Arms: Bausch & Lomb Multi-Purpose Solution
Device: Ciba's Multi-Purpose Solution — Lens care product for disinfecting lenses on a daily basis.
  Arms: Ciba's Multi-Purpose Solution

SUMMARY:
The objective of this study is to evaluate the clinical performance of Bausch & Lomb investigational Multi-Purpose Solution compared to Ciba Vision Multi-Purpose Solution when used by wearers of silicone hydrogel or Group IV contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be of legal age (at least 18) on the date the Informed Consent Form (ICF) is signed and with the capacity to provide voluntary informed consent.
* Participants must habitually use a lens care product for lens cleaning, disinfecting, and storage.
* Participants must wear a lens in each eye and each lens must be of the same manufacture and brand.
* Participants must agree to wear study lenses on a daily wear basis.
* Participants must be able and willing to comply with all treatment and follow-up/study procedures.

Exclusion Criteria:

* Participants participating in any drug or device clinical investigation within 2 weeks prior to entry into this study and/or during the period of study participation.
* Participants with any systemic disease affecting ocular health.
* Participants using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Participants who have had any corneal surgery (eg, refractive surgery).
* Participants who are allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This one month study was conducted at 20 sites by 20 investigators in the United States. First participant was enrolled 11/30/2009 and last Participants visit was 1/22/2010.
Pre-assignment Details: 312 participants(624 eyes) started the study, 7 of which were ineligible at baseline, one was non-dispensed. 305(610 eyes) participants were eligible. 3 participants were discontinued during the study. 302 participants (604 eyes) completed the study.
Period: Enrolled Participants
Arm/Group | Bausch & Lomb Multi-Purpose Solution | Ciba's Multi-Purpose Solution
Started | 156 | 156
Completed | 153 | 152
Not Completed | 3 | 4
Not completed — Ineligible at baseline | 3 | 4
Period: Eligible Participants
Arm/Group | Bausch & Lomb Multi-Purpose Solution | Ciba's Multi-Purpose Solution
Started | 153 | 152
Completed | 153 | 149
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bausch & Lomb Multi-Purpose Solution | Ciba's Multi-Purpose Solution | Total
Number analyzed (Participants) | 153 | 152 | 305
Age, Customized [Number; unit: participants]
  Between 18 and 70 years | 153 | 152 | 305
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 112 | 214
  Male | 51 | 40 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 131 | 126 | 257
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Comfort-related Symptoms/Complaints
Description: Participants rated their subjective symptoms/complaints using a 0 to 100 scale for each eye. A 0 represented the least favorable rating, and a 100 represented the most favorable rating. Over All Follow-Up Visits summarizes the average over all follow-up visit summaries.
Time Frame: At dispensing visit and each follow-up visit at week 2 and week 4.
Population: Summaries included all eligible, dispensed participants, with participants summarized under the study products received.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Multi-Purpose Solution | Ciba's Multi-Purpose Solution
Number analyzed (Participants) | 153 | 151
Number analyzed (eyes) | 306 | 302
Units on a scale
  Comfort | 89.0 (14.2) | 88.3 (14.7)
  End of Day Comfort | 81.7 (20.7) | 81.9 (17.4)
  Burning/stinging upon insertion | 91.4 (15.6) | 93.1 (14.0)
  Irritation | 88.2 (17.1) | 89.3 (14.1)
  Itching | 91.2 (15.8) | 94.3 (10.3)
  Dryness | 84.9 (20.6) | 85.4 (15.8)
  Redness | 90.7 (16.4) | 92.8 (13.0)

2. Secondary Outcome: Slit Lamp Findings
Description: Graded slit lamp findings for each eye greater than grade 2 included epithelial edema, epithelial microcysts, corneal staining, limbal injection, bulbar injection, superior tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates. Slit lamp findings are grade on a scale of 0-4 with 0=none and 4=severe. Over All Follow-up Visits summarizes the worst case over all follow-up visits.
Time Frame: Over all visits for 1 month
Population: Greater than grade 2 for all dispensed eyes with non-missing scores
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Multi-Purpose Solution | Ciba's Multi-Purpose Solution
Number analyzed (Participants) | 156 | 153
Number analyzed (eyes) | 312 | 306
eyes | 1 | 3

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse events measured by eye
Arm/Group | Bausch & Lomb Multi-Purpose Solution | Ciba's Multi-Purpose Solution
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/156
Other Adverse Events (participants affected / at risk) | 0/156 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor.